CLINICAL TRIAL: NCT03242057
Title: Comparison of Primary Extubation Failure Between Non-invasive Positive Pressure Ventilation (NIPPV) and Non Invasive Neural Access Ventilatory Assist (NI-NAVA)
Brief Title: Comparison of Primary Extubation Failure Between NIPPV and NI-NAVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201701971
Record Dates: First submitted 2017-07-28; First posted 2017-08-08 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Preterm Infant; BPD - Bronchopulmonary Dysplasia; Barotrauma
Keywords: NAVA; Extubation; NIPPV
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia; Barotrauma

STUDY DESIGN:
Masking Description: provider and PI is masked for randomization but then no masking once treatment (mode of ventilation) is applied
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NI-NAVA (Experimental): * Wait to meet extubation criteria within 14 days postnatal age
  * Pre-extubation mode of invasive ventilation will be per physician discretion (NAVA, CMV, high frequency oscillator ventilation (HFOV) or high frequency jet ventilation (HFJV)) Pi to determine eligibility or exclusion
  * Randomize to either NIPPV or NI-NAVA, 1:1 randomization
  * PI will not be blinded to the intervention (not feasible)
  * If extubating to NAVA then place the catheter to optimize position and Edi 1 hr. prior to planned extubation.
  * ABG or CBG to be obtained at 4 hrs. post extubation
  * NI-NAVA settings will be weaned or increased as the clinical situation demands and outlined in the protocol
  Interventions: Other: NAVA
- NIPPV (Active Comparator): Wait to meet extubation criteria within 14 days postnatal age
  * Pre-extubation mode of invasive ventilation will be per physician discretion (NAVA, CMV, high frequency oscillator ventilation (HFOV) or high frequency jet ventilation (HFJV)) PI to determine eligibility or exclusion
  * Randomize to either NIPPV or NI-NAVA, 1:1 randomization
  * PI will not be blinded to the intervention (not feasible)
  * ABG or CBG to be obtained at 4 hrs. post extubation
  * NIPPV settings will be weaned or increased as the clinical situation demands and outlined in the protocol
  Interventions: Other: NIPPV

INTERVENTIONS:
Other: NAVA — Infant will be extubated to NAVA, settings based per protocol
  Arms: NI-NAVA
Other: NIPPV — Infant will be extubated to NIPPV, settings detailed in protocol
  Arms: NIPPV

SUMMARY:
Extubation failure is a significant problem in preterm neonates and prolonged intubation is a well-documented risk factor for development of chronic lung disease. Out of the respiratory modalities available to extubate a preterm neonate; high flow nasal canula, nasal continuous positive airway pressure (nCPAP) and noninvasive positive pressure ventilation (NIPPV) are the most commonly used.

A recent Cochrane meta-analysis concluded that NIPPV has lower extubation failure as compared to nCPAP (30% vs. 40%)

NAVA (neurally adjusted ventilatory assist), a relatively new mode of mechanical ventilation in which the diaphragmatic electrical activity initiates a ventilator breath and adjustment of a preset gain (NAVA level) determines the peak inspiratory pressure. It has been reported to improve patient - ventilator synchrony and minimize mean airway pressure and ability to wean an infant from a ventilator. However till date there has been no head to head comparison of extubation failure in infants managed on NAVA with conventional ventilator strategies.

In this study the investigators aim to compare primary extubation failure rates in infants/participants managed by NIPPV vs. NI-NAVA (non invasive NAVA). Eligible infants/participants will be randomized to be extubated to predefined NIPPV or NI-NAVA ventilator settings and will be assessed for primary extubation failure (defined as reintubation within 5 days after an elective extubation).

DETAILED DESCRIPTION:
Mechanical ventilation is needed for most preterm infants to maintain adequate oxygenation and ventilation. However the coexistence of lung immaturity, weak respiratory drive, excessively compliant chest wall, and surfactant deficiency often contribute to dependency on mechanical ventilation during the first days or weeks after birth.

Prolonged mechanical ventilation is associated with high mortality and morbidities including ventilator-associated pneumonia, pneumothorax, and bronchopulmonary dysplasia (BPD). Each additional week of mechanical ventilation is reported to be associated with an increase in the risk of neurodevelopmental impairment. Reduction in the need and duration of invasive mechanical ventilation may potentially improve outcome of preterm infants.

Extubation failure has been independently associated with increased mortality, longer hospitalization, and more days on oxygen and ventilatory support. It is critical, therefore, to attempt extubation early and at a time when successful extubation is likely.

A recent Cochrane review compared the use of nasal intermittent positive pressure ventilation (NIPPV) with nasal continuous positive airway pressure (nCPAP) in preterm infants after extubation and found that NIPPV may be more effective than nCPAP at decreasing extubation failure.

The feasibility of NAVA use has been described in neonatal and pediatric patients. Several studies cite a decrease in peak inspiratory pressures, improved synchrony in triggering, and more appropriate termination of positive pressure support. Some studies have reported lower work of breathing, PaO2/FiO2 ratios (partial pressure of oxygen/ fractional inspired oxygen)and MAP. In addition, NAVA has been used for patients who "fight the ventilator," and the synchrony improves the ability to wean.

The use of NIV-NAVA in neonates has promise as a primary mode of ventilation to aid in the prevention of intubation and also maintaining successful extubation. Early extubation may be enhanced with NIV-NAVA of those neonates requiring intubation for numerous reasons. The ability to provide synchronous NIV allows clinicians the opportunity to extubate infants earlier with increased confidence than with previous post extubation support.

However there is lack of scientific evidence on extubation failure rates on NI-NAVA. Trials comparing NAVA to conventional ventilators with regard to ventilator associated lung injury, ventilator associated pneumonia and decreasing duration of time on the ventilator have not yet been reported.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born between 24 weeks and ≤ 32 weeks completed gestational age or birth weight less than or equal to 1500 grams
2. Postnatal age ≤ 14 days
3. Inborn
4. Mechanically ventilated for at least 12 hrs.
5. Intubated within first 24 hrs. after birth
6. Outborn infants intubated and transferred to UF within 24 hrs. after birth.

Exclusion Criteria:

1. Outborn > 24hrs of age.
2. Failed elective extubation prior to study enrollment
3. Major congenital anomalies or known/suspected chromosomal anomalies
4. Use of paralytics in previous 24 hrs.
5. Participation in another randomized interventional trial
6. Known or suspected phrenic nerve palsy or lesion
7. Known or suspected diaphragmatic lesion
8. Any contraindication to have a nasogastric or orogastric tube placement

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Extubation success | 5 days
  assess how many infants stayed extubated at 5 days after extubation

SECONDARY OUTCOMES:
Bronchopulmonary dysplasia (BPD) | until discharge / 36 weeks post menstrual age
  based on NIH guidelines
Ventilator Days | until discharge / 36 weeks post menstrual age
  days on positive pressure ventilation
NICU length of stay | until discharge / 36 weeks post menstrual age
  discharge or death or transfer
Patent ductus arteriosus (PDA) | until discharge / 36 weeks post menstrual age
  echo diagnosed/confirmed
Necrotizing enterocolitis (NEC | until discharge / 36 weeks post menstrual age
  confirmed on Xray
Late onset sepsis | until discharge / 36 weeks post menstrual age
  only culture proven
Gastrointestinal perforation | until discharge / 36 weeks post menstrual age
  confirmed on X-ray or surgical exploration
Mortality | until discharge / 36 weeks post menstrual age
  all causes within NICU stay
Extubation failure at 3 days | until discharge / 36 weeks post menstrual age
  reintubation by 72 hrs. post extubation
Extubation failure at 7 days | until discharge / 36 weeks post menstrual age
  reintubation by 72 hrs. post extubation
Pulmonary air leak | until discharge / 36 weeks post menstrual age
  including pulmonary interstitial emphysema (PIE) pneumomediastinum and pneumothorax
Severe intraventricular hemorrhage | until discharge / 36 weeks post menstrual age
  on cranial ultrasound, worst grade
Abdominal distension > 2cm from baseline and with signs necessitating cessation of feeds during the first 48 hrs. after extubation | until discharge / 36 weeks post menstrual age
  during the first 48 hrs. after extubation
Retinopathy of prematurity (ROP) | until discharge / 36 weeks post menstrual age
  ophthalmologic exam
Ventilator associated Pneumonia (VAP) | until discharge / 36 weeks post menstrual age
  diagnosed based on tracheal culture + CXR changes + clinical worsening + treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sanket Shah, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Firestone KS, Beck J, Stein H. Neurally Adjusted Ventilatory Assist for Noninvasive Support in Neonates. Clin Perinatol. 2016 Dec;43(4):707-724. doi: 10.1016/j.clp.2016.07.007. PMID 27837754
- [Background] LoVerde B, Firestone KS, Stein HM. Comparing changing neurally adjusted ventilatory assist (NAVA) levels in intubated and recently extubated neonates. J Perinatol. 2016 Dec;36(12):1097-1100. doi: 10.1038/jp.2016.152. Epub 2016 Sep 15. PMID 27629375
- [Background] Firestone KS, Fisher S, Reddy S, White DB, Stein HM. Effect of changing NAVA levels on peak inspiratory pressures and electrical activity of the diaphragm in premature neonates. J Perinatol. 2015 Aug;35(8):612-6. doi: 10.1038/jp.2015.14. Epub 2015 Mar 12. PMID 25764328
- [Background] Stein H, Firestone K. Application of neurally adjusted ventilatory assist in neonates. Semin Fetal Neonatal Med. 2014 Feb;19(1):60-9. doi: 10.1016/j.siny.2013.09.005. Epub 2013 Nov 13. PMID 24238745
- [Background] Stein H, Firestone K, Rimensberger PC. Synchronized mechanical ventilation using electrical activity of the diaphragm in neonates. Clin Perinatol. 2012 Sep;39(3):525-42. doi: 10.1016/j.clp.2012.06.004. PMID 22954267
- [Background] Lemyre B, Davis PG, De Paoli AG, Kirpalani H. Nasal intermittent positive pressure ventilation (NIPPV) versus nasal continuous positive airway pressure (NCPAP) for preterm neonates after extubation. Cochrane Database Syst Rev. 2017 Feb 1;2(2):CD003212. doi: 10.1002/14651858.CD003212.pub3. PMID 28146296
- [Background] Lee J, Kim HS, Jung YH, Shin SH, Choi CW, Kim EK, Kim BI, Choi JH. Non-invasive neurally adjusted ventilatory assist in preterm infants: a randomised phase II crossover trial. Arch Dis Child Fetal Neonatal Ed. 2015 Nov;100(6):F507-13. doi: 10.1136/archdischild-2014-308057. Epub 2015 Jul 15. PMID 26178463
- [Background] Baudin F, Pouyau R, Cour-Andlauer F, Berthiller J, Robert D, Javouhey E. Neurally adjusted ventilator assist (NAVA) reduces asynchrony during non-invasive ventilation for severe bronchiolitis. Pediatr Pulmonol. 2015 Dec;50(12):1320-7. doi: 10.1002/ppul.23139. Epub 2014 Dec 8. PMID 25488197
- [Background] Bhandari V. Nasal intermittent positive pressure ventilation in the newborn: review of literature and evidence-based guidelines. J Perinatol. 2010 Aug;30(8):505-12. doi: 10.1038/jp.2009.165. Epub 2009 Oct 22. PMID 19847188